CLINICAL TRIAL: NCT05824949
Title: The Impact of Osseodensification and Conventional Drilling Protocols on Implants Mechanical and Biological Stability in Posterior Maxilla: A Randomized Controlled Clinical Trial
Brief Title: Osseodensification Versus Conventional Drilling Effect on Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Ta'a, Associate Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Implant stability
Record Dates: First submitted 2023-04-10; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Implant Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseodensification (test) group (Experimental): installation of 40 implants using the osseodensification protocol + measurement of implant stability (ISQ)
  Interventions: Procedure: osseodensification drilling
- Conventional (control) group (Active Comparator): installation of 40 implants using the conventional drilling protocol + measurement of implant stability (ISQ)
  Interventions: Procedure: conventional drilling

INTERVENTIONS:
Procedure: osseodensification drilling — Implant mechanical and biological stability measured using ISQ values at the time of implant placement and at abutment connection for 40 implants placed in the posterior maxillary area using the osseodensification protocol.
  Arms: Osseodensification (test) group
Procedure: conventional drilling — Implant mechanical and biological stability measured using ISQ values at the time of implant placement and at abutment connection for 40 implants placed in the posterior maxillary area using the conventional drilling protocol.
  Arms: Conventional (control) group

SUMMARY:
A total of 80 implants were placed in the posterior region of the maxilla in 40 patients in a split-mouth design. Bone quality was classified into type I, II, III, IV, or V as assessed preoperatively on cone-beam computed tomography (CBCT) . Primary implant stability was measured with insertion torque and resonance frequency analysis (ISQ values). Secondary stability was measured by ISQ at abutment installation.

ELIGIBILITY:
Inclusion Criteria:

* (a) Bilateral edentulism in the maxillary posterior region dating back more than 6 months,
* (b) sufficient bone height (distance between the bone crest and maxillary sinus >8 mm) and width at the alveolar crest (≥6 mm) that would not necessitate bone augmentation,
* (c) at least 2 mm vestibular keratinized mucosa width and 3 mm mucosa thickness,
* (d) full-mouth plaque and bleeding scores <20%.

Exclusion Criteria:

* patients with systemic diseases, conditions, or used medications having the potential to impair surgery, bone, and wound healing dynamics (such as diabetes) will be excluded.
* patients who are allergic to antibiotics and non-steroidal anti-inflammatory drugs
* bone height <8mm
* ridge and soft tissue deficiencies requiring augmentation procedures and
* endodontic or periodontal lesions neighboring the edentulous sites will be also excluded.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Mechanical or primary stability | directly after implant placement
  ISQ values at implant installation
Biological or secondary stability | 4 months after implant installation
  ISQ values at abutment connection

SECONDARY OUTCOMES:
Torque value (N/cm) | directly after implant insertion
  Torque value shown at the physiodispenser screen at the end of implant installation

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Abu-Ta'a, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided